CLINICAL TRIAL: NCT06810648
Title: Effect of Epidural Analgesia on Goal-Directed Fluid Therapy Using Stroke Volume Variation in Elective Major Abdominal Surgery Involving Low Risk Patients: A Cohort Study
Brief Title: Epidural Analgesia and Intraoperative Fluid Management in Colorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Agathi Karakosta, Assistant Professor of Anaesthesiology, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-15/09/2016
Record Dates: First submitted 2025-01-17; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: ERAS; Colorectal Surgery; Goal-directed Fluid Therapy; Conventional Fluid Therapy; Epidural Analgesia

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into four groups based on different anesthetic modalities for intraoperative fluid management and analgesic strategy: The GDFT group received goal-directed fluid therapy and continuous intravenous analgesia, the GDFT/ED group received goal-directed fluid therapy and epidural analgesia, the CFT group received conventional fluid administration and continuous intravenous analgesia, and the CFT/ED group received conventional fluid administration and epidural analgesia. Data for the GDFT and GDFT/ED groups were collected prospectively, while data for the CFT and CFT/ED groups were collected retrospectively
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GDFT group (Experimental): Patients in the GDFT group were managed perioperatively using goal-directed fluid administration and continuous intravenous analgesia.
  Interventions: Procedure: GDFT
- GDFT/ED group (Experimental): Patients in the GDFT/ED group were managed perioperatively using goal-directed fluid administration and epidural analgesia.
  Interventions: Procedure: GDFT/ED
- CFT (Experimental): Patients in the CFT group were managed perioperatively using conventional fluid administration and continuous intravenous analgesia.
  Interventions: Procedure: CFT
- CFT/ED (Experimental): Patients in the CFT group were managed perioperatively using conventional fluid administration and epidural analgesia.
  Interventions: Procedure: CFT/ED

INTERVENTIONS:
Procedure: GDFT — Hydration was goal-directed and guided by Stroke Volume Variation (SVV) using the FloTrac/Vigileo monitor, while analgesia was provided with intravenous analgesics.
  Other Names: Prospective group
  Arms: GDFT group
Procedure: GDFT/ED — Hydration was goal-directed and guided by Stroke Volume Variation (SVV) using the FloTrac/Vigileo monitor, while analgesia was administered via epidural analgesics.
  Other Names: Prospective group
  Arms: GDFT/ED group
Procedure: CFT — Patients received conventional fluid therapy (based on heart rate, urine output and mean arterial pressure) and analgesia was provided with intravenous analgesics.
  Other Names: Retrospective group
  Arms: CFT
Procedure: CFT/ED — Patients received conventional fluid therapy (based on heart rate, urine output and mean arterial pressure) and analgesia was administered via epidural analgesics.
  Other Names: Retrospective group
  Arms: CFT/ED

SUMMARY:
The Enhanced Recovery After Surgery (ERAS) protocols have demonstrated their efficacy in expediting recovery and minimizing postoperative complications, especially in patients undergoing abdominal surgery. Perioperative hydration is one of the most critical pillars of the ERAS protocols, with goal-directed methods for administering fluids increasingly incorporated into these protocols.

The Goal-Directed Fluid Therapy (GDFT) method is a strategy used in perioperative and critical care settings to optimize fluid administration tailored to a patient's individual needs. Its goal is to maintain adequate tissue perfusion and oxygenation by precisely balancing fluid administration, avoiding both hypovolemia (too little fluid) and fluid overload. Rather than using a "one-size-fits-all" approach, GDFT adjusts fluid delivery based on real-time monitoring of the patient's physiological parameters. GDFT focuses on dynamic hemodynamic indicators, such as stroke volume (SV), stroke volume variation (SVV), and cardiac output (CO), which provide better insight into the patient's fluid responsiveness. Advanced monitoring tools, such as esophageal Doppler, pulse contour analysis, or invasive devices like a pulmonary artery catheter, are used to assess the patient's response to fluid administration. The implementation of such protocols, particularly in colorectal surgery, has proven beneficial, as both overhydration and underhydration in this context can significantly impair organ function and, consequently, affect patient outcomes. Hypovolemia may lead to tissue ischemia at the anastomotic site, potentially causing breakdown. Conversely, fluid overload can have harmful consequences; hyperhydration may cause tissue edema, thereby reducing anastomotic strength. However, these findings have been validated primarily in high-risk patients, with a limited number of studies involving low- to moderate-risk patients undergoing major abdominal surgery.

Colorectal surgery is routinely managed with epidural analgesia combined with general anaesthesia. However, concerns have been raised that epidurally induced sympathetic blockade and vasoplegia (vasodilation) can cause haemodynamic instability, necessitating fluid and vasopressor administration to an uncertain extent.

In this single-center trial, we aimed to investigate whether epidural analgesia, in addition to general anaesthesia, influences Stroke Volume Variation (SVV)-guided GDFT using the FloTrac/Vigileo monitor during major open abdominal surgery. The study hypothesis was that epidural analgesia may result in fluid overload to compensate for the induced vasoplegia and that this fluid overload, in turn, could lead to gastrointestinal dysfunction and prolong the length of hospital stay.

The primary outcomes were the incidence of postoperative gastrointestinal dysfunction and the length of hospital stay following elective colorectal surgery in patients managed with GDFT, either with or without epidural analgesia. Additionally, patient records of those treated with conventional fluid therapy (CFT), with or without epidural analgesia, were reviewed retrospectively for comparison.

DETAILED DESCRIPTION:
Existing evidence regarding the implementation of Enhanced Recovery After Surgery (ERAS) protocols highlights their benefits in accelerating the recovery process and reducing hospital stay durations. Additionally, postoperative morbidity, mortality, and rehospitalization rates are lower in patients following these protocols. A key component of ERAS protocols is perioperative fluid management, which is critical for gastrointestinal recovery after major abdominal surgery. Both overhydration and underhydration can significantly impair organ function and, consequently, affect patient outcomes.

Goal-directed fluid therapy (GDFT), utilizing dynamic volume measurements, enables balanced fluid administration. Numerous studies support the implementation of such protocols, particularly in major abdominal surgeries. Colonic anastomotic leakage is one of the most serious complications following colorectal surgery, with a reported incidence of up to 20%. Anastomotic breakdown is associated with increased morbidity and mortality, resulting in prolonged hospitalization, depletion of healthcare resources, and elevated costs. Hypovolemia can lead to tissue ischemia at the anastomotic site, causing breakdown. Conversely, fluid overload may have harmful consequences; hyperhydration can lead to tissue edema, thereby reducing anastomotic strength. These findings underscore the importance of maintaining euvolemia during colorectal surgeries, supporting the inclusion of GDFT as an essential component of the anesthetic protocol. However, the benefits of GDFT in abdominal surgery have been predominantly investigated and validated in high-risk patients. Only a limited number of studies involve low- to moderate-risk patients undergoing major abdominal surgery.

Epidural analgesia, combined with general anaesthesia, is considered the gold standard anaesthetic regimen for major abdominal surgery. However, the resulting sympathetic blockade and vasoplegia can cause haemodynamic instability, affecting fluid administration and vasopressor requirements to an uncertain extent. Various clinical and laboratory markers have been employed to monitor the effects of perioperative fluid management. Evidence suggests that B-type Natriuretic Peptide (BNP) levels are associated with fluid balance, morbidity and mortality at 30 days or even 180 days after non-cardiac surgery, and length of hospital stay. However, the concept of using risk predictors such as BNP in surgeries involving significant fluid loss and redistribution, such as colorectal surgeries, remains insufficiently studied.

This single-center trial was conducted to investigate whether epidural analgesia, in addition to general anaesthesia, influences Stroke Volume Variation (SVV) guided GDFT using the FloTrac/Vigileo monitor in major open abdominal surgery. The study hypothesis was that epidural analgesia may result in overhydration to compensate for the induced vasoplegia, thereby affecting gastrointestinal function and length of hospital stay. The primary outcome was the effect of epidural analgesia on the incidence of postoperative gastrointestinal dysfunction and the length of hospital stay in low- to moderate-risk patients undergoing open major abdominal surgery managed with intraoperative GDFT. Secondary outcomes included the total volume of fluids administered, assessment of proBNP levels as a marker of fluid balance, incidence of postoperative adverse events, and all-cause in-hospital mortality. Additionally, patients' records treated with conventional fluid therapy (CFT) with or without epidural analgesia were reviewed retrospectively for comparison.

ELIGIBILITY:
Inclusion Criteria:

* adults
* elective oncological colorectal surgery
* ASA (American Society of Anesthesiologists physical status classification) I & II

Exclusion Criteria:

* extremes of weight (< 55 kg or > 120 kg)
* known history of arrhythmias
* recent unstable coronary syndrome
* decompensated heart failure
* severe aortic valve stenosis
* impaired renal function (serum creatinine level > 2.0 mg/dL)
* inability to communicate
* refusal to provide consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal dysfunction | From day of surgery untill 30 days after surgery.
  Postoperative ileus, anastomotic leak, anastomotic breakdown, gastrointestinal bleeding.
Length of hospital stay | From day of admission to day of discharge, an average of 30 days.
  Duration (days) from admission to hospital discharge

SECONDARY OUTCOMES:
Total fluids | From beginning of surgery until PACU (post anaesthesia care unit) discharge, an average of 5 hours.
  Total volume of fluids administered intraoperatively.
proBNP levels | From 20-24 hours before surgery to 20-24 hours after surgery.
  Measurement of proBNP (pro B-type natriuretic peptide) blood levels at two time points: pre- and postoperatively.
All-cause in hospital mortality | From day of admission to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Total number of deaths that occur within a hospital setting, regardless of the underlying cause.
Postoperative pulmonary complications | From day of surgery to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Respiratory infection, respiratory failure, pleural effusion, atelectasis, pneumothorax, bronchospasm, aspiration pneumonitis, acute respiratory distress syndrome [ARDS], pulmonary edema, exacerbation of pre-existing lung disease, and pulmonary embolism.
Major adverse cardiovascular events | From day of surgery to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Stroke, myocardial infarction, cardiovascular death
Acute kidney injury | From day of surgery to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Postoperative injury to the kidneys is reflected by at least a twofold increase in baseline serum creatinine.
Reoperation | From day of surgery to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Need for reoperation and return to the theater after PACU (post anaesthesia care unit) discharge.
ICU admission | From day of surgery to day of discharge from the hospital or day of death during hospitalization, whichever comes first, an average of 30 days.
  Unplanned ICU (intensive care medicine) admission after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - "Attikon" Hospital, Athens, Attica
  - University Hospital of Ioannina, Ioannina, Epirus